CLINICAL TRIAL: NCT01775124
Title: A 24-month, Randomized, Double-masked, Controlled, Multicenter Study Evaluating the Efficacy and Safety of Ranibizumab 0.5 mg Administered as Two Alternative Dosing Regimens in Chinese Patients With Neovascular Age Related Macular Degeneration (AMD)
Brief Title: Efficacy and Safety of Ranibizumab 0.5 mg Administered as Two Alternative Dosing Regimens in Chinese Patients With nAMD (Age Related Macular Degeneration)
Acronym: DRAGON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002A2413
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Macular degeneration,; age-related macular degeneration (ARMD),; vision loss,; macula damage,; retina damage,; dry macular degeneration,; wet macular degeneration,; AMD
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 0.5 mg monthly (Experimental): Monthly intravitreal injections of ranibizumab 0.5 mg in the core treatment period and PRN intravitreal injections of the same dose guided by best-corrected visual acuity (BCVA) stabilization in the extension treatment period
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg pro re nata (PRN) (Experimental): PRN intravitreal injections of ranibizumab 0.5 mg guided by best-corrected visual acuity (BCVA) stabilization in the 23 month treatment period
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of 0.5 mg Ranibizumab

SUMMARY:
The study evaluated the efficacy and safety of two different dosing regimens of ranibizumab (either monthly injections or injections as-needed based on the stability of a patient's vision) in Chinese patients with wet age-related macular degeneration (AMD) . This study was to provide long-term safety data in the treatment of Chinese patients with wet AMD.

ELIGIBILITY:
Key Inclusion criteria:

* Patients with visual impairment due to neovascular AMD
* A qualifying vision score at study entry Key Exclusion criteria
* Active infection or inflammation either eye at study entry
* Uncontrolled glaucoma in either eye
* Any disorder in the study eye which may affect vision
* Use of any systemic anti-vascular endothelial growth factor (VEGF)-drugs within 3 months prior to study entry
* Previous treatment of the study eye for wet AMD
* Any surgery in the study eye 3 months prior to or planned with 6 month after study entry

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2015-11-23 (Actual); Study Completion 2015-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- China (17):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 334 patients were randomized in this study. One patient was mis-randomized to ranibizumab 0.5 monthly group and another patient was discontinued due to AE. Neither patient received any treatment
Groups:
- Ranibizumab 0.5 mg Monthly: Monthly intravitreal injections of ranibizumab 0.5 mg in the core treatment period and PRN intravitreal injections of the same dose guided by BCVA stabilization in the extension treatment period
- Ranibizumab 0.5 mg PRN: PRN intravitreal injections of ranibizumab 0.5 mg guided by BCVA stabilization in the 23 month treatment period
Period: Core Period
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Started | 168 | 166
Full Analysis Set | 167 | 166
Per Protocol Set | 157 | 155
Safety Set | 166 (1 patient was mis-randomized & 1 patient discontinued due to AE. No treatment given) | 166
Completed | 157 | 156
Not Completed | 11 | 10
Not completed — Disease Progression | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Death | 0 | 1
Not completed — Administrative problems | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 5 | 5
Period: Extension Period
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Started | 157 | 156
Completed | 145 | 138
Not Completed | 12 | 18
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Administrative problems | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN | Total
Number analyzed (Participants) | 167 | 166 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (8.43) | 66.8 (8.31) | 66.2 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 95
  Male | 119 | 119 | 238

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Visual Acuity (Letters) From Month 3 to Month 4 Through Month 12
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like VA testing charts at a testing distance of 4 meters. This outcome measure describes the difference between the VA averaged across all visits from Month 4 through 12 and the Month 3 Level of Visual Acuity (Letters) of the Study Eye. The treatment regimen up to Month 3 is the same in both treatment groups.
Time Frame: Month 3 to month 4 through Month 12
Population: Full Analysis Set: Consisted of all patients to whom study treatment was assigned. Following the intent to treat principle, patients were analyzed according to the treatment they were assigned to at randomization. (MV-LOCF)=Mean value interpolation and last observation carried forward
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 162 | 159
Letters | 3.3 (5.61) | 1.7 (6.87)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg Monthly vs Ranibizumab 0.5 mg PRN; Descriptive, no hypothesis; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.95 to -0.2]

2. Secondary Outcome: Average Visual Acuity Change (Letters) From Month 3 to Month 4 Through Month 24
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes the difference between the average level of VA over all monthly post-baseline assessments from Month 4 to Month 24 and the Month 3 Level of VA. The treatment regimen up to Month 3 is the same in both treatment groups.
Time Frame: Month 3 to month 4 through Month 24
Population: Full Analysis Set: Consisted of all patients to whom study treatment were assigned. Following the intent to treat principle, patients were analyzed according to the treatment they were assigned to at randomization. (MV-LOCF)=Mean value interpolation and last observation carried forward
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 162 | 159
Letters | 3.7 (7.36) | 2.2 (7.95)

3. Secondary Outcome: Average Visual Acuity Change From Baseline to Month 1 Through Month 12 and Month 1 Through Month 24
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes the difference between VA averaged across all visits from Month 1 through Month 12 (24) and the baseline VA level
Time Frame: Baseline to Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 165 | 166
Letters
  Average Month 1 through month 12 | 10.1 (9.37) | 8.1 (10.95)
  Average Month 1 through month 24 | 11.0 (10.28) | 8.9 (11.95)

4. Secondary Outcome: Change From Baseline in Visual Acuity (Letters) of the Study Eye Over Time
Description: Visual acuity (VA) was assessed on both eyes during every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes the change in visual acuity at each visit compared to baseline
Time Frame: Baseline to 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 165 | 166
letters
  Month 1 | 4.3 (6.75) | 3.4 (8.74)
  Month 2 | 6.8 (8.02) | 6.3 (9.94)
  Month 3 | 8.0 (9.38) | 7.2 (11.48)
  Month 4 | 9.3 (10.52) | 7.9 (11.67)
  Month 5 | 9.9 (10.71) | 8.4 (11.66)
  Month 6 | 10.7 (10.92) | 8.7 (12.33)
  Month 7 | 11.4 (10.49) | 8.5 (13.01)
  Month 8 | 11.3 (11.06) | 8.8 (12.53)
  Month 9 | 11.8 (10.90) | 9.2 (12.83)
  Month 10 | 12.4 (11.24) | 9.4 (12.84)
  Month 11 | 12.5 (10.90) | 9.6 (12.89)
  Month 12 | 12.3 (11.47) | 9.6 (13.06)
  Month 13 | 12.2 (12.04) | 9.9 (12.98)
  Month 14 | 12.1 (12.18) | 10.0 (13.29)
  Month 15 | 12.2 (12.19) | 9.9 (13.56)
  Month 16 | 12.3 (11.59) | 10.0 (13.64)
  Month 17 | 12.1 (11.94) | 10.4 (13.78)
  Month 18 | 11.8 (12.31) | 10.1 (13.25)
  Month 19 | 12.1 (12.43) | 9.8 (14.54)
  Month 20 | 12.1 (12.70) | 9.8 (14.74)
  Month 21 | 11.9 (13.17) | 9.6 (14.73)
  Month 22 | 11.3 (13.19) | 9.5 (15.26)
  Month 23 | 11.5 (13.23) | 9.2 (15.13)
  Month 24 | 11.3 (13.72) | 9.3 (15.48)

5. Secondary Outcome: Number of Patients With a BCVA Improvement of ≥5, ≥10, ≥15, and ≥30 Letters From Baseline to Month 24
Description: Visual acuity (VA) was at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes for each post-baseline month whether or not a patient improved by equal or more than 5, 10, 15,or 30 letters of VA as compared to baseline.
Time Frame: Baseline to Month 24
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 165 | 166
Patients
  Month 1 Gain of >=5 letters | 75 | 65
  Month 1 Gain of >=10 letters | 27 | 31
  Month 1 Gain of >=15 letters | 11 | 17
  Month 1 Gain of >=30 letters | 1 | 1
  Month 2 Gain of >=5 letters | 98 | 95
  Month 2 Gain of >=10 letters | 54 | 48
  Month 2 Gain of >=15 letters | 28 | 32
  Month 2 Gain of >=30 letters | 1 | 1
  Month 3 Gain of >=5 letters | 107 | 100
  Month 3 Gain of >=10 letters | 71 | 60
  Month 3 Gain of >=15 letters | 40 | 37
  Month 3 Gain of >=30 letters | 1 | 4
  Month 4 Gain of >=5 letters | 115 | 100
  Month 4 Gain of >=10 letters | 80 | 75
  Month 4 Gain of >=15 letters | 53 | 46
  Month 4 Gain of >=30 letters | 3 | 4
  Month 5 Gain of >=5 letters | 114 | 109
  Month 5 Gain of >=10 letters | 88 | 72
  Month 5 Gain of >=15 letters | 59 | 46
  Month 5 Gain of >=30 letters | 4 | 5
  Month 6 Gain of >=5 letters | 124 | 108
  Month 6 Gain of >=10 letters | 86 | 75
  Month 6 Gain of >=15 letters | 60 | 44
  Month 6 Gain of >=30 letters | 6 | 9
  Month 7 Gain of >=5 letters | 127 | 114
  Month 7 Gain of >=10 letters | 89 | 70
  Month 7 Gain of >=15 letters | 63 | 50
  Month 7 Gain of >=30 letters | 5 | 10
  Month 8 Gain of >=5 letters | 129 | 110
  Month 8 Gain of >=10 letters | 89 | 74
  Month 8 Gain of >=15 letters | 66 | 54
  Month 8 Gain of >=30 letters | 6 | 7
  Month 9 Gain of >=5 letters | 126 | 107
  Month 9 Gain of >=10 letters | 95 | 78
  Month 9 Gain of >=15 letters | 69 | 57
  Month 9 Gain of >=30 letters | 6 | 11
  Month 10 Gain of >=5 letters | 128 | 116
  Month 10 Gain of >=10 letters | 95 | 75
  Month 10 Gain of >=15 letters | 74 | 53
  Month 10 Gain of >=30 letters | 8 | 11
  Month 11 Gain of >=5 letters | 130 | 115
  Month 11 Gain of >=10 letters | 97 | 77
  Month 11 Gain of >=15 letters | 78 | 56
  Month 11 Gain of >=30 letters | 7 | 11
  Month 12 Gain of >=5 letters | 129 | 114
  Month 12 Gain of >=10 letters | 97 | 82
  Month 12 Gain of >=15 letters | 69 | 52
  Month 12 Gain of >=30 letters | 7 | 11
  Month 13 Gain of >=5 letters | 127 | 118
  Month 13 Gain of >=10 letters | 96 | 92
  Month 13 Gain of >=15 letters | 67 | 56
  Month 13 Gain of >=30 letters | 9 | 11
  Month 14 Gain of >=5 letters | 124 | 117
  Month 14 Gain of >=10 letters | 100 | 88
  Month 14 Gain of >=15 letters | 70 | 65
  Month 14 Gain of >=30 letters | 9 | 13
  Month 15 Gain of >=5 letters | 126 | 112
  Month 15 Gain of >=10 letters | 104 | 84
  Month 15 Gain of >=15 letters | 68 | 62
  Month 15 Gain of >=30 letters | 8 | 13
  Month 16 Gain of >=5 letters | 126 | 114
  Month 16 Gain of >=10 letters | 101 | 87
  Month 16 Gain of >=15 letters | 71 | 62
  Month 16 Gain of >=30 letters | 7 | 11
  Month 17 Gain of >=5 letters | 119 | 116
  Month 17 Gain of >=10 letters | 102 | 87
  Month 17 Gain of >=15 letters | 71 | 62
  Month 17 Gain of >=30 letters | 5 | 12
  Month 18 Gain of >=5 letters | 121 | 117
  Month 18 Gain of >=10 letters | 101 | 87
  Month 18 Gain of >=15 letters | 69 | 61
  Month 18 Gain of >=30 letters | 6 | 13
  Month 19 Gain of >=5 letters | 121 | 115
  Month 19 Gain of >=10 letters | 94 | 88
  Month 19 Gain of >=15 letters | 75 | 62
  Month 19 Gain of >=30 letters | 9 | 11
  Month 20 Gain of >=5 letters | 116 | 116
  Month 20 Gain of >=10 letters | 98 | 85
  Month 20 Gain of >=15 letters | 72 | 63
  Month 20 Gain of >=30 letters | 10 | 13
  Month 21 Gain of >=5 letters | 120 | 117
  Month 21 Gain of >=10 letters | 96 | 81
  Month 21 Gain of >=15 letters | 76 | 61
  Month 21 Gain of >=30 letters | 11 | 12
  Month 22 Gain of >=5 letters | 116 | 114
  Month 22 Gain of >=10 letters | 92 | 88
  Month 22 Gain of >=15 letters | 69 | 64
  Month 22 Gain of >=30 letters | 14 | 13
  Month 23 Gain of >=5 letters | 119 | 115
  Month 23 Gain of >=10 letters | 93 | 85
  Month 23 Gain of >=15 letters | 72 | 62
  Month 23 Gain of >=30 letters | 8 | 13
  Month 24 Gain of >=5 letters | 114 | 116
  Month 24 Gain of >=10 letters | 95 | 83
  Month 24 Gain of >=15 letters | 73 | 60
  Month 24 Gain of >=30 letters | 11 | 13

6. Secondary Outcome: Number of Patients With a BCVA Loss of 15 Letters in the Study Eye Over Time
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes for each post-baseline month whether or not a patient lost less than 15 letters of VA as compared with baseline.
Time Frame: Baseline to Month 24
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 165 | 166
Patients
  Month 1, Loss of < 15 letters | 164 | 163
  Month 2, Loss of < 15 letters | 163 | 162
  Month 3, Loss of < 15 letters | 160 | 162
  Month 4, Loss of < 15 letters | 161 | 162
  Month 5, Loss of < 15 letters | 160 | 160
  Month 6, Loss of < 15 letters | 162 | 160
  Month 7, Loss of < 15 letters | 162 | 158
  Month 8, Loss of < 15 letters | 162 | 159
  Month 9, Loss of < 15 letters | 163 | 159
  Month 10, Loss of < 15 letters | 162 | 161
  Month 11, Loss of < 15 letters | 162 | 161
  Month 12, Loss of < 15 letters | 162 | 160
  Month 13, Loss of < 15 letters | 162 | 157
  Month 14, Loss of < 15 letters | 161 | 158
  Month 15, Loss of < 15 letters | 162 | 159
  Month 16, Loss of < 15 letters | 163 | 159
  Month 17, Loss of < 15 letters | 161 | 157
  Month 18, Loss of < 15 letters | 159 | 157
  Month 19, Loss of < 15 letters | 162 | 155
  Month 20, Loss of < 15 letters | 161 | 155
  Month 21, Loss of < 15 letters | 157 | 155
  Month 22, Loss of < 15 letters | 160 | 154
  Month 23, Loss of < 15 letters | 158 | 153
  Month 24, Loss of < 15 letters | 158 | 153

7. Secondary Outcome: Number of Patients With a Best Corrected Visual Acuity (BCVA) of More of 73 Letters or More
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes for Month 12 and Month 24 whether a patient had a VA score of 73 or more letters
Time Frame: Month 12 and 24
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 165 | 166
Patients
  Month 12>=73 letters | 68 | 56
  Month 24>=73 letters | 63 | 59

8. Secondary Outcome: Change From Baseline in Central Sub-Field Thickness (CSFT) of the Study Eye Over Time to Month 12 and Month 24
Description: Optical coherence tomography(OCT) was used to assess CSFT (Central Sub-Field Thickness) representing the average retinal thickness of the circular area within 1 mm diameter around the foveal center. The Ns in the rows is the number of patients with a value for both baseline and the specific post-baseline visit
Time Frame: Baseline to Month 24
Population: Full Analysis Set: Consisted of all patients to whom study treatment were assigned. Following the intent to treat principle, patients were analyzed according to the treatment they were assigned to at randomization. (LOCF)= last observation carried forward
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 163 | 166
microns
  Month 1 | -112.8 (117.95) | -108.7 (124.93)
  Month 2 | -141.1 (126.44) | -130.4 (145.58)
  Month 3 | -141.3 (127.47) | -141.2 (161.88)
  Month 4 | -150.4 (131.71) | -134.5 (158.88)
  Month 5 | -155.2 (134.58) | -131.5 (155.98)
  Month 6 | -158.6 (135.37) | -138.3 (159.07)
  Month 7 | -156.9 (136.61) | -137.9 (165.24)
  Month 8 | -165.4 (135.59) | -142.2 (165.76)
  Month 9 | -165.1 (136.04) | -143.3 (176.68)
  Month 10 | -165.9 (136.03) | -152.5 (177.11)
  Month 11 | -166.6 (140.62) | -152.5 (175.56)
  Month 12 | -166.5 (143.85) | -155.7 (173.19)
  Month 13 | -160.3 (142.02) | -151.4 (168.89)
  Month 14 | -159.9 (144.14) | -153.2 (167.81)
  Month 15 | -156.9 (152.33) | -158.1 (169.56)
  Month 16 | -155.9 (154.82) | -158.1 (173.23)
  Month 17 | -161.8 (155.18) | -156.8 (167.89)
  Month 18 | -159.5 (159.78) | -156.7 (174.88)
  Month 19 | -158.5 (163.82) | -154.8 (177.49)
  Month 20 | -157.6 (161.04) | -152.1 (173.30)
  Month 21 | -155.2 (160.03) | -151.9 (171.95)
  Month 22 | -156.8 (161.35) | -146.5 (176.83)
  Month 23 | -159.4 (163.58) | -148.3 (185.62)
  Month 24 | -167.7 (163.12) | -153.2 (178.22)

9. Secondary Outcome: Duration of Ranibizumab Treatment Free Interval in the Study Eye up to Month 24
Description: This outcome measure describes duration of treatment-free intervals. Treatment-free interval is defined as the number of visits (whether attended or not) where ranibizumab was not administered. n= the number of patients who had at least one ranibizumab treatment interruption
Time Frame: up to month 24
Population: Safety set consisted of all patients who received at least one application of ranibizumab ( active study treatment) and had at least one post-baseline safety assessment. A patient who had no AEs also constituted a safety assessment
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 166 | 166
Months
  First treatment free interval (n=99,144) | 2.9 (2.38) | 3.7 (4.67)
  Second treatment free interval (n=49,112) | 2.1 (1.51) | 3.3 (3.48)
  Third treatment free interval (n=12,78) | 1.5 (0.52) | 3.0 (2.67)

10. Secondary Outcome: Duration of Ranibizumab Treatment Free Interval in the Study Eye Prior to Month 12
Description: This outcome measure describes duration of treatment-free intervals prior to month 12. Treatment-free interval is defined as the number of visits (whether attended or not) where ranibizumab was not administered. n= the number of patients who had at least one ranibizumab treatment interruption Treatment-free interval is analyzed in the Ranibizumab 0.5 mg PRN group only. It is not analyzed in the Ranibizumab 0.5 mg monthly group because, by protocol design, these participants receive treatment monthly. Therefore, the analysis does not apply to this group.
Time Frame: prior to month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 166
Months
  First treatment free interval (n=127) | 2.7 (2.22)
  Second treatment free interval (n=73) | 2.0 (1.29)
  Third treatment free interval (n=19) | 1.3 (0.67)

11. Secondary Outcome: Duration of Active Treatment Phase Prior to Month 12
Time Frame: Prior to month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 166 | 166
Months | 10.5 (1.86) | 9.1 (2.76)

12. Secondary Outcome: Duration of Active Treatment Phase up to Month 24
Time Frame: up to month 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Number analyzed (Participants) | 166 | 166
Months | 18.0 (5.99) | 17.1 (6.90)

ADVERSE EVENTS:
Description: Safety Set: consisted of all patients who received at least one application of ranibizumab (the active study treatment) and had at least one post-Baseline safety assessment. A patient who had no AEs also constituted a safety assessment.
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 0.5 mg PRN
Serious Adverse Events (participants affected / at risk) | 24/166 | 24/166
Other Adverse Events (participants affected / at risk) | 107/166 | 87/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly (N=166) | Ranibizumab 0.5 mg PRN (N=166)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 4 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly (N=166) | Ranibizumab 0.5 mg PRN (N=166)
Cardiac discomfort (Cardiac disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Age-related macular degeneration (Eye disorders) | 3 | 1
Cataract (Eye disorders) | 2 | 2
Choroidal neovascularisation (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 21 | 12
Conjunctival hyperaemia (Eye disorders) | 1 | 2
Conjunctivitis allergic (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 2 | 2
Eye pain (Eye disorders) | 4 | 1
Foreign body sensation in eyes (Eye disorders) | 4 | 3
Glaucoma (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 4 | 1
Macular fibrosis (Eye disorders) | 1 | 2
Macular oedema (Eye disorders) | 0 | 4
Neovascular age-related macular degeneration (Eye disorders) | 1 | 2
Ocular hyperaemia (Eye disorders) | 2 | 1
Retinal haemorrhage (Eye disorders) | 5 | 6
Retinal tear (Eye disorders) | 1 | 2
Vision blurred (Eye disorders) | 1 | 3
Visual acuity reduced (Eye disorders) | 7 | 2
Vitreous detachment (Eye disorders) | 1 | 2
Chronic gastritis (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 6 | 5
Malaise (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 5 | 3
Herpes zoster (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 24 | 18
Pneumonia (Infections and infestations) | 2 | 1
Pulpitis dental (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 7
Urinary tract infection (Infections and infestations) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 2 | 0
Blood glucose increased (Investigations) | 10 | 5
Blood pressure increased (Investigations) | 1 | 3
Blood uric acid increased (Investigations) | 4 | 5
Intraocular pressure increased (Investigations) | 5 | 12
Visual acuity tests abnormal (Investigations) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 5 | 7
Headache (Nervous system disorders) | 3 | 2
Lacunar infarction (Nervous system disorders) | 0 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary.

However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety